CLINICAL TRIAL: NCT01858610
Title: Drug Interaction Between Irbesartan and Hydrochlorothiazide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damanhour University (Other)
Responsible Party: Principal Investigator, Sally Helmy, PhD, CPHQ, Lecturer of Pharmaceutics, Faculty of Pharmacy, Damanhour University
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: PPT4
Record Dates: First submitted 2013-05-12; First posted 2013-05-21 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: Healthy
Keywords: Fixed dose combination; Pharmacokinetics; Irbesartan; Hydrochlorothiazide; Pharmacodynamics; Normotensive Participants
MeSH Terms: interventions — Hydrochlorothiazide; Irbesartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Irbesartan alone (Other): Irbesartan 300 mg alone
  Interventions: Drug: Irbesartan
- Hydrochlorothiazide 25 mg alone (Other): Hydrochlorothiazide 25 mg alone
  Interventions: Drug: Hydrochlorothiazide
- Irbesartan 300 mg + Hydrochlorothiazide 25 mg (Other): Irbesartan 300 mg + Hydrochlorothiazide 25 fixed dose combination
  Interventions: Drug: Irbeasartan/hydrochlorothiazide

INTERVENTIONS:
Drug: Irbeasartan/hydrochlorothiazide
  Other Names: Fixed dose combination
  Arms: Irbesartan 300 mg + Hydrochlorothiazide 25 mg
Drug: Irbesartan
  Arms: Irbesartan alone
Drug: Hydrochlorothiazide
  Arms: Hydrochlorothiazide 25 mg alone

SUMMARY:
This study was conducted to investigate any potential reaction between irbesartan and hydrochlorothiazide.

ELIGIBILITY:
Inclusion Criteria:

At least 18 years old and not more than 45 healthy normotensive male volunteers Who had passed all the screening parameters

Exclusion Criteria:

A clinically significant abnormal physical exam, medical history, or laboratory studies If they showed a sitting SBP of >140 or <100 mmHg, DBP > 90 or <60mm Hg, or a pulse rate of > 95 or < 50 beats/min at screening The use of any prescription drug within the previous month or use of any over-the-counter medication within the past 14 days A history of blood dyscrasias A history of alcohol or drug abuse within the past year Donation of blood during the 8 weeks prior to the study or plans to donate blood during or within 8 weeks of completing the study Unable to tolerate vein puncture and multiple blood samplings Any surgical/medical condition that might alter drug absorption, distribution, metabolism, or excretion

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2013-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Blood pressure (systolic/diastolic) | participants will be followed for the duration of hospital stay, an expected average of 5 weeks
pharmacokinetic parameter such as the Cmax of irbesartan and hydrochlorothiazide | After collection of all blood samples, an expected average of 4 weeks
Heart rate | participants will be followed for the duration of hospital stay, an expected average of 5 weeks
pharmacokinetic parameter such as the AUC of irbesartan and hydrochlorothiazide | After collection of all blood samples, an expected average of 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmaceutics Department, Faculty of Pharmacy, Damanhour University, Damanhur, Egypt

REFERENCES:
- [Derived] Hedaya MA, Helmy SA. Modeling of the pharmacokinetic/pharmacodynamic interaction between irbesartan and hydrochlorothiazide in normotensive subjects. Biopharm Drug Dispos. 2015 May;36(4):216-31. doi: 10.1002/bdd.1935. Epub 2015 Feb 4. PMID 25545238